CLINICAL TRIAL: NCT04539145
Title: Chocolate PTA Balloon Compared to Conventional Balloon Angioplasty for Sustained Lumen Gain in Below the Knee Arteries - CHOCO-CABANA Trial-
Brief Title: CHOCO-CABANA Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klinikum Rosenheim (Other)
Collaborators: Medtronic (Industry); Herz-Zentrums Bad Krozingen (Other); University Hospital Tuebingen (Other); Klinikum Karlsbad-Langensteinbach (Other); Elblandklinikum Radebeul Interdisziplinäres Gefäßzentrum Radebeul / Riesa (Unknown); LKH-Universitätsklinikum Graz Univ. Klinik für Innere Medizin Klin. Abteilung für Angiologie (Unknown); Hanusch-Krankenhaus Kardiovaskuläres Zentrum (Unknown); Auckland City Hospital (Other Government); SCO:SSiS (Unknown); coreLab Black Forest GmbH (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Gunnar Tepe, Chief Physician of the Radiology Department, Klinikum Rosenheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RO-012020
Record Dates: First submitted 2020-08-04; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: 120 patients (60 per group) Special balloon (chocolate balloon with a special nitiol cage around the balloon - not drug coated) versus standard uncoated balloon
Who Masked: Participant
Masking Description: Randomization per envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chocolate PTA balloon (Experimental)
  Interventions: Device: Chocolate PTA Balloon
- POBA (Other): Intervention with regular baloon
  Interventions: Device: conventional balloon angioplasty

INTERVENTIONS:
Device: Chocolate PTA Balloon — Chocolate PTA Balloon
  Arms: Chocolate PTA balloon
Device: conventional balloon angioplasty — conventional bal-loon angioplasty
  Arms: POBA

SUMMARY:
The study will be performed 120 patients at about 6 to 8 study centers. Only patients with clinical conditions requiring assessment of patency of the treated BTK lesions at 6 months post procedure by MRA as part of standard care to prevent amputations as consequence of non-detected re-stenosis/occlusions will be included in the study. The sequence in which the individual patients will be treated will be randomized with the Chocolate PTA balloon and the uncoated conventional PTA balloon at each center. 60 patients will be randomized to uncoated conventional PTA balloon treatment and 60 patients to treatment with the Chocolate PTA balloon.

All lesions in each patient (lesions that fulfill the inclusion/exclusion criteria) should be treated as the patient is randomized.

In patients with long lesions more than one balloon may be used. Overlapping of balloons (at least 10mm) is mandatory to avoid untreated gaps between sequential treatments. Follow up will be performed at 1 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Chronic stenotic or occlusive atherosclerotic disease of the infrapopliteal arteries
3. Patients with clinical conditions requiring assessment of vessel patency of treated BTK lesion 6 months post procedure as part of clinical standard of care to prevent amputa-tions as consequence of non-detected re-stenosis
4. BTK intervention with lesions between 1 and 25 cm
5. Sufficient outflow of the treated artery to the foot (less than 50% stenosis or sufficient collaterals)
6. All BTK lesions either to be treated with conventional PTA or with the Chocolate PTA balloon (if inclusion criteria 4 and 5 apply)*

   * The longest lesion will be taken as primary lesion. All other lesions will be also analyzed within the study protocol but separately evaluated. If a secondary lesion does not fulfill the inclusion criteria 4 and 5, the lesion can be treated upon the decision of the operator and will not be analyzed within the study protocol.
7. Rutherford 3-5 patients
8. Patients who are able to be followed to assess vessel patency according to standard lo-cal hospital care (e.g. DUS, MRA)
9. Successfully treated inflow lesions up to TASC B

Exclusion Criteria:

1. Acute or sub-acute thrombosis
2. In-stent restenosis
3. Rutherford 1-2 and 6
4. Patient who is not fit for follow-up (including contraindication for MRA)
5. Vessel preparation with cutting balloon, lithotripsie, atherectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-03-27 (Estimated); Study Completion 2022-03-27 (Estimated)

PRIMARY OUTCOMES:
Recoil (lumen loss > 30%) 15-30 min after study intervention angiographically documented and analyzed by a core-lab | 15-30 min after study intervention
  The minimal lumen of the artery in the area of Intervention in mm will be compared directly after the Intervention and at 15-30 minuntes

SECONDARY OUTCOMES:
the loss of patency greater than 50% in the MRA after six month | 6 month
  the lumen of the artery directly after the Intervention, 15 min after the Intervention and at 6 months will be compared (in mm). It is a secondary outcome if the loss is greater than 50%
the re-occlusion rate at 6 months (measured by MRA) | 6 month
  lumen = 0 mm = recocclusion
Residual stenosis (MLD post compared to RVD, % of RVD) >50% after the invention | immedetely after the intervention
  interventional success: lumen of the artery directly after the Intervention (compared to the healthy vessel next to the lesion - in mm) - RVD = reference vessel Diameter, MLD = Minimum lumen diameter
Wound status at 1 and 6 months: | 1 and 6 months
  as estimated by the patient (healed, improved, no change, worsened)
target lesion revascularization TLR rate at 1 and 6 months | 1 and 6 months
  if an endovascular of surgical therapy of the lesion which was treated is performed
Amputation rate at 1 and 6 months | 1 and 6 months
Clinical presentation (Rutherford 0, 1, 2, 3, 4, 5 or 6 at 30 days and 6 months | 1 and 6 month
  Rutherford 0 = no symptoms, Rutherford 6 = worst symptoms
Ancle brachial index (ABI) compared to baseline and post intervention and 6 months | directly after the intervention and 6 month
  Blood pressure in the arm divided by blood pressure in the distal leg (normal value: 0.8-1.2)
DUS vs. MRA at 6 months | 6 month
  both by DUS and MRA % Stenosis of the index lesion will be calculated. They will be compared in order to see if DUS has the same value as MRA

CONTACTS AND LOCATIONS:
Locations (8):
- Austria (2):
  - LKH-Univ. Klinikum Graz, Graz
  - Hanusch-Krankenhaus Kardiovaskuläres Zentrum, Vienna
- Germany (5):
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad (Baden), Baden-Wuettenberg
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Tepe, Rosenheim, Baden-Wurttemberg
  - Uniklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Elblandklinikum Radebeul Interdisziplinäres Gefäßzentrum Radebeul / Riesa, Radebeul
- Auckland City Hospital, Grafton, New Zealand